CLINICAL TRIAL: NCT01576991
Title: Telomeres and Reproduction in Women
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 108093
Record Dates: First submitted 2012-04-10; First posted 2012-04-13 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: InVitro Fertilization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Follicle cells, and or polar body of eggs
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Oocyte collection: This is an observational study; there are no cohorts or groups

SUMMARY:
The purpose of the study is to describe the relationship between leukocyte, granulose cell and polar body telomere length, telomere injury foci (TIFs), polarized light microscopy of oocyte spindles and their frequency in the eggs from older women and associations with aneuploidy.

DETAILED DESCRIPTION:
The chances of conception decrease and miscarriage increase with a women's age, and the locus of reproductive aging is the egg (1). Egg dysfunction affects most women beginning by their late '30's and for many women age related egg dysfunction represents a major cause of infertility. The cause of age related egg dysfunction is poorly understood, but telomere dysfunction may play an important role. Our group has demonstrated that genetic or pharmacologic shortening of telomeres in the eggs of mice, which normally do not exhibit age related egg dysfunction, mimics reproductive aging in women, with cell cycle arrest, apoptosis, spindle dysmorphologies and chromosomal abnormalities (1,2). Moreover, a pilot study the investigators conducted five years ago suggested that telomere length of spare human eggs may predict the outcome of womens' InVitro Fertilization (IVF) cycles (3). Subsequently, other investigators have demonstrated that telomere length of circulating leukocytes predicts miscarriages (4).

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 48
* Undergoing InVitro Fertilization
* Willing to donate spare eggs, granulosa cells and blood
* Willing to give written informed consent

Exclusion Criteria:

* Not undergoing InVitro Fertilization
* Not willing to donate spare eggs, granulosa cells or blood
* Not willing to give written informed consent
* Previously donated spare eggs, granulosa cells or blood for this research project

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: InVItro Fertilization patients undergoing therapy
Sampling Method: Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2009-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Telomere length | 1 year
  Describe the relationship between leukocyte, granulose cell and polar body telomere length, telomere injury foci (TIFs), polarized light microscopy of oocyte spindles

SECONDARY OUTCOMES:
Frequency of telomeres | 1 year
  The Primary outcome frequencies in the eggs from older women and associations with aneuploidy.

CONTACTS AND LOCATIONS:
Overall Officials: Celso Silva, MD, Principal Investigator — University of South Florida